CLINICAL TRIAL: NCT04325932
Title: Study of Urinary Kallikrein to Enhance Collateral Circulation in Symptomatic Intracranial Atherosclerosis: a Study Based on Whole-brain CTP
Brief Title: Study of Urinary Kallikrein to Enhance Collateral Circulation in Symptomatic Intracranial Atherosclerosis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UK-001
Record Dates: First submitted 2017-10-05; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2015-05

CONDITIONS: Intracranial Arteriosclerosis; Collateral Circulation; Anterior Cerebral Circulation Infarction
MeSH Terms: conditions — Intracranial Arteriosclerosis; Brain Infarction | interventions — Tissue Kallikreins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Urinary Kallikrein group (Experimental): Urinary Kallikrein for injection, 0.15PNA IU,qd, for 2 weeks, administered within 96 hours after TIA or acute ischemic stroke, with basic therapies like dual antiplatelet therapy, blood pressure-lowering therapy and lipid-lowering therapy.
  Interventions: Drug: Urinary Kallikrein
- control group (No Intervention): with basic therapies like dual antiplatelet therapy, blood pressure-lowering therapy and lipid-lowering therapy.

INTERVENTIONS:
Drug: Urinary Kallikrein
  Other Names: Urinary Kallidinogenase
  Arms: Urinary Kallikrein group

SUMMARY:
The purpose of this study is to determine whether Urinary Kallikrein has an additional effect on enhancing collateral circulation in symptomatic intracranial atherosclerotic patients under clopidogrel and aspirin dual antiplatelet therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke or TIA within 72 hours;
2. Intracranial ICA, MCA M1 segment stenosis (>70%)

Exclusion Criteria:

1. >70% Stenosis in an intracranial artery other than the culprit artery.
2. >50% Stenosis of an extracranial carotid or vertebral artery on the ipsilateral side.
3. Perforator strokes based on MRI.
4. Non-atherosclerotic lesion, for example, moyamoya disease, vascular inflammatory disease due to infection, autoimmunity diseases, developmental or genetic abnormalities, for example, fibromuscular dysplasia, sickle-cell anaemia, suspected vasospasm.
5. Potential cardiac embolism as cause.
6. Intracranial haemorrhage within 6 weeks.
7. Concomitant intracranial tumour, aneurysm or arteriovenous malformation.
8. Known contraindications for heparin, aspirin, clopidogrel or contrast.
9. Haemoglobin <10 g/dL, blood platelet count <100 000, international normalisation ratio >1.5, or other uncorrectable coagulopathies.Impaired liver function (alanine aminotransferase or glutamic oxalacetic transaminase ≥ 3×upper limit of normal) or renal function (serum creatinie ≥ 1.5mg/dl);
10. A baseline modified Rankin Score of ≥3.
11. Life expectancy of <1 year due to the concomitant illness.
12. Pregnant or lactating women.
13. long-term statins users.
14. History of mental instability or dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
the percentage of patients with modified Rankin Score (mRS) equivalent to or less than 2 | 3 months

SECONDARY OUTCOMES:
rLMC scale of Collateral circulation | 2 weeks, 1 month
  We use regional leptomeningeal score(rLMC) score to measure collateral circulation.rLMC score is based on scoring pial and lenticulostriate arteries in 6 ASPECTS regions(M1-6) plus anterior cerebral artery region and basal ganglia. Pial arteries in the Sylvian sulcus are scored 0,2, or 4.
NIHSS score | 2 weeks, 1month
Hemorrhageic complications | 2 weeks, 1 month, 3 months, 6 months
  Hemorrhageic complications including intracranial, digestive tract
New stroke or transient ischemic attack(TIA) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Min Lou, Ph.D,M.D., Study Chair — second affiliated hospital of Zhejiang University, school of medicine
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No